CLINICAL TRIAL: NCT00147459
Title: Immunogenicity of Booster Hepatitis B Vaccines in Children After Liver Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 931205
Record Dates: First submitted 2005-09-05; First posted 2005-09-07 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Liver Transplantation; Hepatitis B
Keywords: hepatitis B virus; vaccine; booster; liver transplantation
MeSH Terms: conditions — Hepatitis B

ARMS (1):
- booster (Active Comparator): no antibody and boosted
  Interventions: Biological: HBV vaccine booster

INTERVENTIONS:
Biological: HBV vaccine booster

SUMMARY:
Aim/Background: This study aims to investigate the necessity and efficacy of a hepatitis B virus (HBV) vaccine booster in children after liver transplantation. A universal mass vaccination program of HBV was launched for 20 years in Taiwan. The coverage rate is high and the effect is great. The carrier rate of the population under vaccine coverage decreased from 10-15% to < 1%. In Taiwan, most children who receive organ transplantation were vaccinated with HBV vaccine in infancy and well before the transplantation procedure. This vaccination background information on Taiwanese children is quite unique and not similar to the other countries in the world. The antibody generated by the vaccine usually wanes after a certain period even in normal subjects, let alone in subjects who receive organ transplantation and immunosuppressive agents after transplantation. At present, Taiwan is still an HBV hyperendemic area and the risk of exposure to HBV cannot be overlooked. Should children be given a booster dose of HBV vaccine after transplantation? And how about the immunogenicity of this booster dose in these immunocompromised hosts? If these children cannot obtain an adequate antibody titer, will the risk of HBV infection increase? This study is designed to answer these questions. As a pediatric hepatologist, the author's routine work is to take care of children who underwent liver transplantation. To take advantage of this, the investigators decided to study the efficacy and necessity of HBV booster vaccine in these patients. However, the results of this study should be able to be applied to any kind of solid organ transplanted patients.

Method: The anti-hepatitis B surface antigen (HBs) titer will be checked in patients who received liver transplantation > 1 year ago. If the titer is < 10 IU/L, a booster dose will be administered. The humoral (anti-HBs) and cellular immunity (by ELISPOT to assay T and B cell specific proliferation) and cytokine assay will be done in these patients before and after the booster dose. A three-year follow-up will be performed to monitor the HBV infection in these patients.

Expected Results: The investigators expect for those who survive one year more after liver transplantation to yield a relatively good response to HBV booster under adequate immunosuppression.

DETAILED DESCRIPTION:
The anti-HBs titer will be checked in the patients who received liver transplantation for > 1 year. If the titer is < 10 IU/L, a booster dose will be administered. The humoral (anti-HBs) and cellular immunity (by ELISPOT to assay T and B cell specific proliferation) and cytokine assay will be done in these patients before and after the booster dose. A three-year follow-up will be performed to monitor the HBV infection in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Children who received liver transplantation > 1 year ago

Exclusion Criteria:

* Are now in an unstable condition

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2005-09; Primary Completion 2006-12 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Persistence of anti-HBs in those primarily vaccinated and who underwent liver transplantation | 1 year
  antibody(+)

SECONDARY OUTCOMES:
The necessity of a booster dose of HBV vaccine for those primarily vaccinated and who underwent liver transplantation | 1 year
  if no antibody , booster

CONTACTS AND LOCATIONS:
Overall Officials: Yen H Ni, MD, PhD, Principal Investigator — NTUH
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan